CLINICAL TRIAL: NCT02084784
Title: Study of Surgical Navigation System in Detection of Sentinel Lymph Node of Early Breast Cancer Patients
Brief Title: Application of Surgical Navigation System in Sentinel Lymph Node of Breast Cancer Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Chinese PLA General Hospital (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Wannan Medical College Yijishan Hospital (Other)
Responsible Party: Principal Investigator, Chongwei Chi, Ph.D, Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011CB707700; 973 (Other Grant/Funding Number: 2011CB707700)
Record Dates: First submitted 2014-03-08; First posted 2014-03-12 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Sentinel Lymph Node; Breast Cancer
Keywords: Near-infrared fluorescence; Image guided surgery; Breast cancer;; Sentinel lymph node biopsy; Indocyanine green; Methylene blue
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indocyanine green & methylene blue, (Experimental): Subcutaneous injection around the areola with 2-4 points Methylene blue with 1ml of 1% Indocyanine green with 1ml of 0.5%
  Interventions: Drug: Indocyanine green; Drug: methylene blue

INTERVENTIONS:
Drug: Indocyanine green — Subcutaneous injection around the areola with 2-4 points Indocyanine green with 1ml of 0.5%
  Other Names: ICG
Drug: methylene blue — Subcutaneous injection around the areola with 2-4 points Methylene blue with 1ml of 1%
  Other Names: MB

SUMMARY:
The purpose of this study is to compare the sentinel lymph node (SLN) detection rate of early breast cancer patients between using Indocyanine green (ICG) and Methylene blue with a novel surgical navigation system.

DETAILED DESCRIPTION:
Assessment of the sentinel lymph node (SLN) in patients with early stage breast cancer is vital in selecting the appropriate surgical approach. However, the existing methods, including methylene blue and nuclides, possess low efficiency and effectiveness in mapping SLNs, and to a certain extent exert side effects during application. Indocyanine green (ICG), as a fluorescent dye, has been proved reliable usage in SLN detection by several other groups. In this paper, the investigators introduce a novel surgical navigation system to detect SLN with ICG. This system contains two charge-coupled devices (CCD) to simultaneously capture real-time color and fluorescent video images through two different bands. During surgery, surgeons only need to follow the fluorescence display. In addition, the system saves data automatically during surgery enabling surgeons to find the registration point easily according to image recognition algorithms. The investigators aim to show that the usage of our surgical navigation system with ICG to detect SLNs in breast cancer patients is technically feasible.

ELIGIBILITY:
Inclusion criteria: (Before the test, all the subjects required for meeting the entry requirements before they join the group)

* female patients;
* The preoperative core needle biopsy or open surgical excision biopsy diagnosis as breast cancer;
* tumor diameter ≤ 3cm;
* No clinical examination of suspicious axillary lymph node-positive;
* diagnosed clinical conditions can be directly surgery as I, II breast cancer patients;
* preoperative clinical or radiologic evidence without distant metastases (M0);
* signed informed consent.

Exclusion criteria: (Before the test, the subjects under any one of items to meet the requirements can not be enrolled)

* Sentinel lymph node biopsy history had received surgery or axillary area;
* multi-center breast cancer or multiple lesions;
* clinical axillary lymph node metastasis have been found;
* mammary area had received neoadjuvant chemotherapy or radiotherapy;
* inflammatory breast cancer;
* pregnancy;
* no personal freedom and independent civil capacity.

Exclusion criteria: (trials, subjects necessary to meet the requirements of any one item, exit the clinical trial research.)

* severe allergic reaction occurs;
* persistent allergic reaction;
* subjects were required to withdraw from a clinical trial;
* researchers consider it not appropriate to continue to participate in the clinical trial investigator.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sentinel lymph node detection rate | 1 year
  Participants will be followed for the duration of hospital stay, an expected average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chongwei Chi, doctor, Study Director — Chinese Academy of Sciences
Locations (1):
- Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Chi C, Ye J, Ding H, He D, Huang W, Zhang GJ, Tian J. Use of indocyanine green for detecting the sentinel lymph node in breast cancer patients: from preclinical evaluation to clinical validation. PLoS One. 2013 Dec 16;8(12):e83927. doi: 10.1371/journal.pone.0083927. eCollection 2013. PMID 24358319
- [Derived] He K, Zhou J, Yang F, Chi C, Li H, Mao Y, Hui B, Wang K, Tian J, Wang J. Near-infrared Intraoperative Imaging of Thoracic Sympathetic Nerves: From Preclinical Study to Clinical Trial. Theranostics. 2018 Jan 1;8(2):304-313. doi: 10.7150/thno.22369. eCollection 2018. PMID 29290809
- [Derived] He K, Chi C, Kou D, Huang W, Wu J, Wang Y, He L, Ye J, Mao Y, Zhang GJ, Wang J, Tian J. Comparison between the indocyanine green fluorescence and blue dye methods for sentinel lymph node biopsy using novel fluorescence image-guided resection equipment in different types of hospitals. Transl Res. 2016 Dec;178:74-80. doi: 10.1016/j.trsl.2016.07.010. Epub 2016 Jul 18. PMID 27497181
- See also: A Website from Key Laboratory of Molecular Imaging, Chinese Academy of Sciences — http://www.mitk.net/